CLINICAL TRIAL: NCT03611972
Title: Effects of Sucrose-sweetened Beverage in African-American and Caucasian Women.
Brief Title: Sucrose-sweetened Beverage in African-American and Caucasian Women.
Acronym: SAAC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI resigned
Sponsor: University of California, Davis (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Office of Research on Women's Health (ORWH) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1243331; K12HD051958 (NIH); UL1TR001860 (NIH)
Record Dates: First submitted 2018-07-27; First posted 2018-08-02 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Healthy
MeSH Terms: interventions — Sugar-Sweetened Beverages

STUDY DESIGN:
Intervention Model Description: Dietary intervention
Masking Description: All outcomes measures are analyzed using only the participant's study ID number.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sugar-sweetened beverage (SSB) (Experimental): SSB provided at 25% of daily energy requirement Frequency: Divided into 3 servings/day Duration: 2 weeks
  Interventions: Dietary Supplement: Sugar-sweetened beverage

INTERVENTIONS:
Dietary Supplement: Sugar-sweetened beverage — Sugar-sweetened koolaid-flavored water.

SUMMARY:
The main objective of this pilot study is to measure changes in metabolic risk factors of cardiovascular disease and type 2 diabetes in response to sugar-sweetened beverages in African-American and non-Hispanic white women.

DETAILED DESCRIPTION:
This is a dietary intervention during which participants will consume a SSB daily, with each meal for two weeks. At the beginning and end of the two-week intervention, participants will have blood drawn under fasting and postprandial (after a meal) conditions for the measurement of lipid risk factors associated with cardiovascular disease. Participants will also undergo an oral glucose tolerance test (OGTT) to assess insulin sensitivity. All sugar-sweetened beverages will be provided.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25 - 35 kg/m2

Exclusion Criteria:

* Does not identify as African-American or non-hispanic White
* Glucose intolerance (fasting glucose >100 mg/dl)
* Evidence of liver disorder (AST or ALT >200% upper limit of normal range)
* Evidence of kidney disorder (>2.0mg/dl creatinine)
* Evidence of thyroid disorder (out of normal range)
* Systolic blood pressure consistently over 140mmHg or diastolic blood pressure over 90mmHg
* Triglycerides > 150mg/dl
* LDL-C > 130mg/dl
* Hemoglobin < 8.5 g/dL
* Pregnant or lactating women
* Current, prior (within 12 months), or anticipated use of any hypolipidemic or anti-diabetic agents PROTOCOL TITLE: The Effects of Sucrose Beverage on African-American and Caucasian Women (SAAC) Study Page 4 of 18 Revised: November 27, 2013
* Use of thyroid, anti-hypertensive, anti-depressant, weight loss medications or any other medication which, in the opinion of the investigator, may confound study results
* Use of chronic corticosteroids (everyday use for a month or longer)
* Use of tobacco
* Strenuous exerciser (>3.5 hours/week at a level more vigorous than walking)
* Surgery for weight loss
* Diet exclusions: Food allergies, special dietary restrictions, food allergies, routine consumption of less than 3 meals/day, routine ingestion of more than 2 sugar-sweetened beverages or 1 alcoholic beverage/day, unwillingness to consume any food on study menu
* Veins that are assessed by the CCRC R.N.s as being unsuitable for long-term infusions and multiple blood draws from a catheter
* Any other condition that, in the opinion of the investigators, would put the subject at risk
* We will exclude individuals from each of the following special populations:

  * Adults unable to consent
  * Individuals who are not yet adults (infants, children, teenagers < 18 years)
  * Pregnant women
  * Prisoners

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 9 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Triglycerides | 2 weeks
  Fasting and postprandial plasma triglycerides
Total cholesterol | 2 weeks
  Fasting and postprandial plasma cholesterol
Low-density lipoprotein (LDL) | 2 weeks
  Fasting and postprandial plasma low-density lipoprotein (LDL)
Oral glucose tolerance test (OGTT) | 2 weeks
  Participants will drink a beverage containing 75g of glucose and blood will be drawn before the drink and at 30 minutes, 60 minutes, 90 minutes, 120 minutes and 180 minutes after the drink. Plasma glucose and insulin will be measured at each time point.

SECONDARY OUTCOMES:
Waist circumference | 2 weeks
  Waist circumference

CONTACTS AND LOCATIONS:
Overall Officials: Candice Price, PhD, Principal Investigator — University of California, Davis
Locations (2):
- United States (2):
  - University of California, Davis, Davis, California
  - University of California, Davis CTSC Clinical Research Center, Sacramento, California

REFERENCES:
- See also: Learn more or sign up for the study here! — https://studypages.com/s/the-effects-of-sucrose-sweetened-beverage-in-african-american-and-caucasian-women-saac-study-734555/